CLINICAL TRIAL: NCT02435719
Title: Effectiveness Evaluation of Alcohol Hand Gel Use in Mbale Regional Referral Hospital, Rural Eastern Uganda
Brief Title: Alcohol Hand Gel Use in Mbale Regional Referral Hospital: a Cost Effectiveness Evaluation
Acronym: WardGel
Status: Completed | Type: Observational
Sponsor: Sanyu Africa Research Institute (Other)
Collaborators: Mbale Regional Referral Hospital (Other); University of Liverpool (Other); Nagasaki University (Other)
Responsible Party: Sponsor
Other Study IDs: SAfRI/OBS/001
Record Dates: First submitted 2015-04-20; First posted 2015-05-06 (Estimated); Last update posted 2016-10-13 (Estimated); Status verified 2016-10

CONDITIONS: Infections, Hospital
Keywords: HCAIs; Handgel; Hospital; Effectiveness
MeSH Terms: conditions — Cross Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Ministry of Health through the National Medical Stores has supplied alcohol-based handgels to the different health facilities in Uganda for the health care providers to use during clinical care. However, constant stock-outs and or limited supplies remains the main constraint faced by the hospitals. Thus the handgels are generally used by a few of the senior health care providers.

The promotion of bedside, antiseptic handrubs largely contributes to the increase in compliance and sustained improvement of hand hygiene compliance reduces Health care acquired infections (HCAIs), but it is not yet established how cost- effective the intervention is in a a rural Ugandan hospital where funds are severely rationed and, which serves over 4 million people in over 15 districts in Uganda. An evaluation of an intervention's cost-effectiveness is a crucial factor in whether the government will be prepared to fund the intervention and sustain it.

This WardGel study thus aims to assess the cost-benefit of providing hand gel for all health care workers in Mbale Regional Referral Hospital.

DETAILED DESCRIPTION:
The WardGel Study aims to assess the cost- effectiveness of providing handgel for all health care workers in selected wards of Mbale regional Referral Hospital in rural Eastern Uganda.

The WardGel study seeks to address the following specific objectives:-

1. To determine the incidence of new infections following hospital admission among in-patients
2. To assess the hand hygiene compliance among the health care providers (HCPs) as the usual practice and with handgel
3. To determine the effectiveness of handgel in reduction of new infections after hospital admission
4. To determine the additional costs associated with development of new infections after hospital stay

This study will compare infection rates before (pre-intervention phase) and after implementation of the hand gel for use by health care providers (intervention phase). The study will also assess hand-hygiene compliance amongst health workers and additional costs associated with management of new acquired infections amongst inpatients while at the hospital.

The pre-intervention phase lasting for 12 weeks will involve baseline evaluation of the current hand hygiene practices on each of the study wards, ascertaining how frequently HCPs washed their hands or used handgel.

At the end of 12 weeks, the Intervention will begin and last for 12 weeks. Alcohol-based hand gels will be introduced and provided to health care providers (HCPs) for use before and after each patient care episode.

In ward Training will be provided for all HCPs, including student trainees of clinical medicine and nursing prior to introduction of the hand gels on its use and any promotion messages for example, displaying posters in each hand washing area in the respective wards. Any other training will be arranged and conducted accordingly. 1-Litre handgel bottles will be fitted in the holders fixed to the walls on the wards, and other free bottles placed on the trolleys for using while conducting ward rounds, others on the reception area during the registration of inpatient, and treatment area while administering patients' treatment.

Also 40ml hand-sized bottles will be availed to health care providers. Additional stocks of the hand gel will be available in the staff areas and one central pharmacy area. Compliance with the intervention will be assessed by direct observation by the research assistants on each ward based on the WHO assessment tools and by volume of gel use.

In both phases, the following will be crosscutting: -

* The study shall adopt the WHO hand hygiene tools (the WHO 5-Moment Tool and hand hygiene compliance tool) to assess the hand hygiene compliance (WHO 2009).
* Prospective data will also be collected daily from all recruited inpatients on the wards prior to and during the implementation of the intervention to document the frequency of infections on admission and the rate of new acquired infections during their hospital stay.

The new infections definitions acquired after admission of the patients and applied in this WardGel study have been developed and modified from the CDC/NHSN Surveillance definitions for specific infections [CDC 2014].

* Individual patients data collected from patient interviews will be augmented by a review of their case files.
* Research assistants will interview all recruited patients and or their carers diagnosed with a new infection to assess the exact extra care costs incurred from patients' perspective. Meanwhile, hospital records shall help to establish the extra costs incurred for antibiotics, and health workers extra time. Other costs will be related hand gel supplies, training and start-up costs.

ELIGIBILITY:
Inclusion Criteria:

* Patients is admitted for at least 24 hours
* Any health care provider, including students

Exclusion Criteria:

* Patients discharged before 24 hours

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will include in-patients and health care providers on six (6) selected wards (Labour ward, Postnatal ward, Gynaecological ward, Acute Care unit, paediatric Ward, and general surgical wards) The sample will be selected by convenience non-probability sampling method
Sampling Method: Non-Probability Sample
Enrollment: 3626 (Actual)
Dates: Start 2014-10; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Evidence of Hospital acquired infection confirmed clinically | At least 48 hours after hospital admission or re-admission.Participants will be followed for the duration of hospital stay, an expected average of 5 days.
  Hospital acquired infection will be defined as new clinically diagnosed infection developed whilst an inpatient or within 2 days of discharge (for readmitted patients).

SECONDARY OUTCOMES:
Evidence of Hospital Acquired infection confirmed by laboratory investigations (CBC and C&S) | At least 48 hours after admission or readmission.Participants will be followed for the duration of hospital stay, an expected average of 5 days.
  Participants will be followed for the duration of hospital stay, an expected average of 5 days.
Hand hygiene compliance by health care providers based on the WHO's 5-moments of Hand hygiene | during patient clinical care.participants will be observed during their clinical care practice, an expected average of 30 minutes per session
  participants will be observed during their clinical care practice, an expected average of 30 minutes per session
cost-effectiveness of hand gel use by micro-economic assessment | Additional period due to confirmed hospital acquired infection.Participants will be followed for the duration of hospital stay, an expected average of 5 days.
  Participants will be followed for the duration of hospital stay, an expected average of 5 days.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Weeks, PhD, Principal Investigator — University of Liverpool; James Ditai, MPH, Principal Investigator — Sanyu Africa Research Institute; Benon Wanume, MMED (CP), Principal Investigator — Mbale Regional Referral Hospital; Julian Abeso, MMED (Paed), Study Director — Mbale Regional Referral Hospital; Kyoko Inoue, MPH, Study Director — Nagasaki University
Locations (1):
- Mbale Regional Referral hospital, Mbale, Uganda

REFERENCES:
- [Derived] Saito H, Inoue K, Ditai J, Wanume B, Abeso J, Balyejussa J, Weeks A. Alcohol-based hand rub and incidence of healthcare associated infections in a rural regional referral and teaching hospital in Uganda ('WardGel' study). Antimicrob Resist Infect Control. 2017 Dec 28;6:129. doi: 10.1186/s13756-017-0287-8. eCollection 2017. PMID 29299303